CLINICAL TRIAL: NCT06772779
Title: A Clinical Study to Evaluate the Effect of MK-0616 on Warfarin and Lisinopril Pharmacokinetics in Healthy Adult Participants
Brief Title: A Study of Enlicitide Decanoate (MK-0616), Warfarin, and Lisinopril in Healthy Adult Participants (MK-0616-026)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-026; MK-0616-026 (Other: MSD)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Warfarin; Vitamin B 6; MK-0616; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Warfarin Plus Enlicitide Decanoate (Experimental): Participants receive oral warfarin and oral enlicitide decanoate.
  Interventions: Drug: Warfarin; Drug: Enlicitide Decanoate
- Lisinopril Plus Enlicitide Decanoate (Experimental): Participants receive oral lisinopril and oral enlicitide decanoate.
  Interventions: Drug: Enlicitide Decanoate; Drug: Lisinopril

INTERVENTIONS:
Drug: Warfarin — single oral dose
  Other Names: Jantoven
  Arms: Warfarin Plus Enlicitide Decanoate
Drug: Enlicitide Decanoate — single oral dose
  Other Names: MK-0616
Drug: Lisinopril — single oral dose
  Other Names: Zestril
  Arms: Lisinopril Plus Enlicitide Decanoate

SUMMARY:
The main goal of this study is to learn what happens in a person's body over time when they take enlicitide decanoate with warfarin or lisinopril. Researchers want to learn if the amount of warfarin in a person's blood is similar when warfarin is taken alone or with enlicitide decanoate.

Enlicitide decanoate is a new medicine that lowers the amount of cholesterol in a person's blood. Warfarin is a drug that reduces risk of blood clotting, and lisinopril is a drug that lowers blood pressure.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to:

* Is in good health
* Has a body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2

Exclusion Criteria:

The key exclusion criteria include but are not limited to:

* History of gastrointestinal disease which may affect food or drug absorption, or has had a gastric bypass or similar surgery
* History of cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the AUC0-Inf of warfarin.
Area Under the Concentration-Time Curve from Time 0 to Last Measurable Concentration (AUC0-Last) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the AUC0-Last of warfarin.
Maximum Plasma Concentration (Cmax) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Cmax of warfarin.
Time to Maximum Plasma Concentration (Tmax) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Tmax of warfarin.
Apparent Terminal Half-life (t½) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the t½ of warfarin.
Apparent Clearance (CL/F) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the CL/F of warfarin.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Warfarin | At designated timepoints (up to approximately 2 weeks postdose)
  Blood samples will be collected to determine the Vz/F of warfarin.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the AUC0-Inf of lisinopril.
Area Under the Concentration-Time Curve from Time 0 to Last Measurable Concentration (AUC0-Last) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the AUC0-Last of lisinopril.
Maximum Plasma Concentration (Cmax) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the Cmax of lisinopril.
Time to Maximum Plasma Concentration (Tmax) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the Tmax of lisinopril.
Apparent Terminal Half-life (t½) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the t½ of lisinopril.
Apparent Clearance (CL/F) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the CL/F of lisinopril.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Lisinopril | At designated timepoints (up to approximately 3 days postdose)
  Blood samples will be collected to determine the Vz/F of lisinopril.

SECONDARY OUTCOMES:
Number of Participants Who Experience a Treatment-Emergent Adverse Event (TEAE) in Part 1 | Up to approximately 5 weeks
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. The number of participants who experience a TEAE in Part 1 will be reported.
Number of Participants Who Discontinue Study due to a TEAE in Part 1 | Up to approximately 5 weeks
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. The number of participants who discontinue study due to a TEAE in Part 1 will be reported.
Number of Participants Who Experience a Treatment-Emergent Adverse Event (TEAE) in Part 2 | Up to approximately 28 days
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. The number of participants who experience a TEAE in Part 2 will be reported.
Number of Participants Who Discontinue Study due to a TEAE in Part 2 | Up to approximately 28 days
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. The number of participants who discontinue study due to a TEAE in Part 2 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com